CLINICAL TRIAL: NCT06076863
Title: Pharmacist Management of Paxlovid eVisits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RDO KPNC 23-096
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Quality of Care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants who review charts will be masked to patient group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist Care (Experimental): Pharmacists on a regional team will manage requests for Paxlovid placed by patients via e-visits using a standard protocol.
  Interventions: Other: Pharmacist Care
- Adult and Family Medicine Physician Pool Care (Active Comparator): Adult and family medicine physicians serving in pools will manage requests for Paxlovid placed by patients via e-visits using a standard protocol.
  Interventions: Other: AFM Pool Care

INTERVENTIONS:
Other: Pharmacist Care — Management of Paxlovid e-visits per regional protocol
  Arms: Pharmacist Care
Other: AFM Pool Care — Management of Paxlovid e-visits per regional and local protocols
  Arms: Adult and Family Medicine Physician Pool Care

SUMMARY:
The goal of this cluster randomized trial is to compare two modes of management -- pharmacist care vs. pooled adult and family medicine physician care -- for electronically submitted requests (e-visits) for Paxlovid by adults with COVID-19. It will compare quality of care based on counseling for common potential drug-drug interactions and time to prescription, as well as the time and financial costs of care in the two groups.

DETAILED DESCRIPTION:
Importance. Enhancing the management of messages from patients and providing virtual options for urgent care are top priorities for The Permanente Medical Group (TPMG) and Kaiser Foundation Hospitals/Health Plan (KFH/P).

Objective. To compare pharmacist management of e-visit requests for Paxlovid for COVID-19 with management by adult and family medicine physician pools regarding costs, time, clinical outcomes, and patient and clinician satisfaction.

Design, setting, and participants. This cluster randomized clinical trial will include adults from 17 medical facilities of Kaiser Permanente Northern California who make Paxlovid e-visits on weekdays from October 9 to December 11, 2023.

Intervention. In the intervention group, a regional team of pharmacists will manage Paxlovid e-visits following a standard protocol; in the comparison group, adult and family medicine physicians (AFMs) will manage these visits according to medical center-based protocols.

Main Outcomes and Measures. The primary outcome is whether a patient with one or more common drug-drug interactions received counseling for any drug-drug interaction. Secondary outcomes are the hours from the e-visit request to the prescription among patients who receive one and the clinician time and cost per visit managed.

Potential Results. We will test the hypotheses that Pharmacist Care compared with AFM Pool Care will have higher quality of care and lower costs based on the receipt of counseling for common drug-drug interactions, faster time to prescriptions, and lower clinician time and cost per visit managed.

Potential Conclusions and Relevance. If pharmacist management has better or similar outcomes compared with AFM pool management, this will provide support to continue this practice for Paxlovid e-visits and to evaluate possible expansion of pharmacist management for similar clinical situations.

ELIGIBILITY:
Inclusion Criteria:

* Patients making Paxlovid e-visits on weekdays from 8:00 am to 4:30 pm during the study period

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2478 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Percent of patients with common potential drug-drug interactions with Paxlovid who received counseling | Within 2 days after the e-visit
  Whether or not a patient with one or more common potential drug-drug interactions with Paxlovid received counseling, as documented in the electronic health record, with data collected via review of text extracts from the EHR

SECONDARY OUTCOMES:
Mean hours from e-visit to Paxlovid prescription, among patients who received one | Within 2 days after the e-visit
  Hours from e-visit to Paxlovid prescription, among patients who received one, measured via analysis of computerized data
Mean minutes of clinician time per Paxlovid e-visit managed | Within 2 days after the e-visit
  Clinician time in minutes per Paxlovid e-visit managed, measured via analysis of computerized data
Personnel cost per Paxlovid e-visit managed | Within 5 days after the e-visit
  Personnel cost per Paxlovid e-visit managed

OTHER OUTCOMES:
Percent of patients rating the quality of care for the Paxlovid e-visit as Excellent or Very Good | At 14 to 28 days after the e-visit
  Patient rating of the quality of care for the Paxlovid e-visit, measured on a 5-point scale with the response options Excelllent, Very Good, Good, Fair, or Poor, with survey responses collected via mail, online, and telephone interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Lieu, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT06076863/Prot_SAP_002.pdf